CLINICAL TRIAL: NCT02894385
Title: A Phase I, Non-randomized, Open-label, Single-dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of BAY 1841788 (ODM-201) in Male Subjects With Hepatic Impairment, Renal Impairment and Normal Hepatic and Renal Function
Brief Title: Effect of Hepatic and Renal Impairment on the Pharmacokinetics, Safety and Tolerability of BAY1841788 (ODM-201)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17721; 2016-001069-10 (EudraCT Number)
Record Dates: First submitted 2016-08-29; First posted 2016-09-09 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Pharmacokinetics; Hepatic Insufficiency; Renal Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 - Subjects with severe renal impairment (Experimental): Subjects with severe renal impairment received a single oral dose of darolutamide 600 mg (2 x 300 mg tablets).
  Interventions: Drug: BAY1841788
- Part 1 - Subjects with moderate hepatic impairment (Experimental): Subjects with moderate hepatic impairment received a single oral dose of darolutamide 600 mg (2 x 300 mg tablets).
  Interventions: Drug: BAY1841788
- Part 1 - Healthy subjects (Experimental): Healthy subjects received a single oral dose of darolutamide 600 mg (2 x 300 mg tablets).
  Interventions: Drug: BAY1841788

INTERVENTIONS:
Drug: BAY1841788 — 600 mg single dose, administered as 2 x 300 mg tablets on Day 00.

SUMMARY:
Evaluate the potential effect of hepatic or renal impairment on the pharmacokinetics, safety and tolerability of BAY 1841788 (ODM-201).

DETAILED DESCRIPTION:
The study was closed after Part 1 because additional investigation in volunteers with moderate renal impairment in Part 2 was not deemed to be ethically or scientifically justified.

ELIGIBILITY:
Inclusion Criteria:

* All subjects

  -- Male and white subjects between 45 and 79 years of age with a body mass index between 18 to 34 kg/m*2 (both inclusive).
* Patients with moderate hepatic impairment (Part 1)

  -- Patients with documented liver cirrhosis confirmed by histopathology, e.g., previous liver biopsy, laparoscopy, ultrasound, or fibroscan and with moderate hepatic impairment (defined as Child Pugh class B).
* Patients with severe renal impairment (Part 1)

  -- Patients with severe renal impairment with an estimated glomerular filtration rate 15-29 mL/min/1.73 m*2, who are not on dialysis and are not expected to start dialysis in the next 3 months (Stage 4).
* Healthy subjects

  -- Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring and with estimated glomerular filtration rate >90 mL/min (according to Modified Diet of Renal Disease equation).
* Patients with moderate renal impairment (Part 2)

  -- Patients with moderate renal impairment with an estimated glomerular filtration rate 30-59 mL/min/1.73 m*2 (Stage 3).
* Patients with mild renal impairment (Part 2)

  -- Patients with mild renal impairment with an estimated glomerular filtration rate (eGFR) 60-79 mL/min/1.73 m*2 (Stage 2).
* Patients with mild hepatic impairment (Part 2)

  * Patients with documented liver cirrhosis confirmed by histopathology, e.g., previous liver biopsy, laparoscopy, ultrasound, or fibroscan.
  * Patients with mild hepatic impairment (defined as Child Pugh class A).

Exclusion Criteria:

* Severe cerebrovascular or cardiac disorders, e.g., myocardial infarction less than 6 months prior to dosing, congestive heart failure of New York Heart Association (NYHA) grade III or IV.
* Subjects with percutaneous transluminal coronary angioplasty or coronary artery bypass graft less than 6 months prior to study drug administration.
* Strong cytochrome P450 (CYP) 3A4 inhibitors or strong CYP3A4 inducers within 28 days or 5 drug half-lives (if drug half-life in patients is known), before start of study treatment.
* Known BCRP (breast cancer resistant protein) and OATP (organic anion-transporting polypeptide) substrates not specifically mentioned in the protocol within 28 days or 5 drug half-lives (if drug half-life in patients is known), before start of study treatment.
* Smoking more than 20 cigarettes daily.

Ages: 45 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of darolutamide from time zero to 48 hours (AUC(0-48)) in plasma | Pre-dose up to 48 h post dose
Maximum drug concentration (Cmax) of darolutamide in plasma | Pre-dose up to 48 h post dose

SECONDARY OUTCOMES:
Area under the concentration-time curve of darolutamide's diastereomer ((S,R)-darolutamide) from time zero to 48 hours (AUC(0-48)) in plasma | Pre-dose up to 48 h post dose
Maximum drug concentration (Cmax) of darolutamide's diastereomer ((S,R)-darolutamide) in plasma | Pre-dose up to 48 h post dose
Area under the concentration-time curve of darolutamide's diastereomer ((S,S)-darolutamide) from time zero to 48 hours (AUC(0-48)) in plasma | Pre-dose up to 48 h post dose
Maximum drug concentration (Cmax) of darolutamide's diastereomer ((S,S)-darolutamide) in plasma | Pre-dose up to 48 h post dose
Area under the concentration-time curve of darolutamide's major metabolite (keto-darolutamide) from time zero to 48 hours (AUC(0-48)) in plasma | Pre-dose up to 48 h post dose
Maximum drug concentration (Cmax) of darolutamide's major metabolite (keto-darolutamide) in plasma | Pre-dose up to 48 h post dose
Number of subjects with study drug-related treatment-emergent adverse events (TEAEs) | From first application of study medication up to 30 days after end of treatment with study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - Kiel, Schleswig-Holstein
  - Lübeck

REFERENCES:
- [Derived] Zurth C, Nykanen P, Wilkinson G, Taavitsainen P, Vuorela A, Huang F, Reschke S, Koskinen M. Clinical Pharmacokinetics of the Androgen Receptor Inhibitor Darolutamide in Healthy Subjects and Patients with Hepatic or Renal Impairment. Clin Pharmacokinet. 2022 Apr;61(4):565-575. doi: 10.1007/s40262-021-01078-y. Epub 2021 Dec 6. PMID 34866168
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/